CLINICAL TRIAL: NCT00390507
Title: Modification of Posttetanic Count (PTC) for Monitoring Deep Neuromuscular Block II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PTC-II
Record Dates: First submitted 2006-10-19; First posted 2006-10-20 (Estimated); Last update posted 2010-09-06 (Estimated); Status verified 2010-09

CONDITIONS: Neuromuscular Blockade
Keywords: Acceleromyography; TOF-Watch; Posttetanic count; Train of four; Neuromuscular blockade

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Post-tetanic count frequency

SUMMARY:
The purpose of this study is to examine the relationship between post-tetanic count (PTC) and time to first response to Train of four (TOF) stimulation during deep neuromuscular blockade induced by rocuronium.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* General anaesthesia >1 hour
* Surgery in supine position with possibility of monitoring the neuromuscular blockade at the thumb (n.ulnaris stimulation).
* Written informed content

Exclusion Criteria:

* Neuromuscular disorders, hepatic and renal dysfunction
* Medication expected to interfere with the neuromuscular blocking agent
* Allergy to any medication used during anaesthesia
* Body weight less or exceeding 20% of the ideal body weight
* Pregnancy or breastfeeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2006-10; Primary Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time to first response to TOF stimulation (T1)

SECONDARY OUTCOMES:
Time to second response to TOF stimulation (T2)
Time to first post-tetanic count (PTC)
Number of post-tetanic count at first response to TOF
Time to T1=25%
Interval 25-75%
Time to TOF 0.9
Time to TOF 1.0

CONTACTS AND LOCATIONS:
Overall Officials: Casper C Kjaer, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (2):
- Denmark (2):
  - Dep. of Anesthesia, Rigshospitalet, Copenhagen, Copenhagen
  - Dep. of Anesthesia, Herlev hospital, Herlev, Herlev